CLINICAL TRIAL: NCT05475886
Title: 6% Hydroxyethyl Starch (130/0.4) Coload for Postspinal Anesthesia Hypotension in Patients Undergoing Caesarean Section: A Randomized Sequential Allocation Dose-finding Study
Brief Title: 6% Hydroxyethyl Starch (130/0.4) Coload for Postspinal Anesthesia Hypotension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Yi Chen-2022-2
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Adverse Effect
Keywords: Hydroxyethyl starch 130/0.4; Coload; Hypotension; Cesarean section
MeSH Terms: conditions — Hypotension | interventions — Hydroxyethyl Starch Derivatives; Colloids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydroxyethyl starch (130/0.4) coload group (Experimental): An initial infusion dose of 500 ml 6% Hydroxyethyl starch (130/0.4) coload simultaneous with spinal anesthesia.
  Interventions: Drug: Hydroxyethyl starch 130/0.4

INTERVENTIONS:
Drug: Hydroxyethyl starch 130/0.4 — An initial infusion dose of 500 ml 6% Hydroxyethyl starch (130/0.4) coload simultaneous with spinal anesthesia. The dose administered to subsequent patients varied by increments or decrements of 100 ml according to the responses of previous patients according to the up-down sequential allocation.
  Other Names: Colloid

SUMMARY:
The purpose of this study is to investigate the ED50 and ED90 for an effective 6% Hydroxyethyl starch (130/0.4) coload infusion dose for postspinal anesthesia hypotension in patients undergoing cesarean section.

DETAILED DESCRIPTION:
Post-spinal anesthesia hypotension is a frequent complication during spinal anesthesia for cesarean section. The incidence of post-spinal anesthesia hypotension is as high as 62.1-89.7% if prophylactic measures are not taken. Colloid fluid coload has been highly demonstrated for prevention and/or treatment of post-spinal anesthesia hypotension. However, the ED50 and ED90 for an effective 6% Hydroxyethyl starch (130/0.4) coload infusion dose for postspinal anesthesia hypotension are still unknown. The purpose of this study is to investigate the ED50 and ED90 for an effective 6% Hydroxyethyl starch (130/0.4) coload infusion dose for postspinal anesthesia hypotension in patients undergoing cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years
* Primipara or multipara
* Singleton pregnancy ≥ 37 weeks
* American Society of Anesthesiologists physical status classification I to II
* Scheduled for elective cesarean section under spinal anesthesia

Exclusion Criteria:

* Body height < 150 cm
* Body weight > 100 kg or body mass index (BMI) ≥ 40 kg/m2
* Eclampsia or chronic hypertension or baseline blood pressure ≥ 160mmHg
* Hemoglobin < 7g/dl
* Coagulation or renal function disorders
* Known allergy to hydroxyethyl starch
* Fetal distress, or known fetal developmental anomaly

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-21 (Estimated); Study Completion 2024-04-21 (Estimated)

PRIMARY OUTCOMES:
ED 50 and ED 90 | 1-15 minutes after spinal anesthesia
  The dose of 6% Hydroxyethyl starch (130/0.4) that would be effective in preventing postspinal anesthesia hypotension in 50% (effective dose, ED 50) and 90% (ED90) of patients

SECONDARY OUTCOMES:
The incidence of post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 80% of the baseline
The incidence of severe post-spinal anesthesia hypotension. | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 60% of the baseline.
The incidence of bradycardia. | 1-15 minutes after spinal anesthesia
  Heart rate < 60 beats/min.
The incidence of nausea and vomiting. | 1-15 minutes after spinal anesthesia
  Presence of nausea and vomiting in patients after spinal anesthesia
The incidence of hypertension. | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) >120% of the baseline.
pH | Immediately after delivery
  From umbilical arterial blood gases.
Partial pressure of oxygen (PO2) | Immediately after delivery
  From umbilical arterial blood gases.
Base excess (BE) | Immediately after delivery
  From umbilical arterial blood gases.
APGAR score | 1 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration
APGAR score | 5 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration

CONTACTS AND LOCATIONS:
Overall Officials: Yi Chen, M.D., Study Chair — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No